CLINICAL TRIAL: NCT03340545
Title: Evaluating Changes in Mechanical Properties in the Herniated Intervertebral Disc
Brief Title: MR Elastography for the Herniated Intervertebral Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Daniel Cortes, Assistant Professor, Penn State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00007840
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-01

CONDITIONS: Intervertebral Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Individuals (Other): Healthy individuals will be imaged for comparison purposes
  Interventions: Other: Custom Magnetic Resonance Elastography Device
- Disc Herniation (Other): Subjects diagnosed with Intervertebral Disc Herniation will be imaged to evaluate sensitivity of the proposed method.
  Interventions: Other: Custom Magnetic Resonance Elastography Device

INTERVENTIONS:
Other: Custom Magnetic Resonance Elastography Device — Magnetic Resonance Elastography is an imaging method to measure mechanical properties of tissues.

SUMMARY:
Low back pain is a major cause of disability, especially in the working-age population. A total of 149 million working days are lost every year as a consequence of back pain. Intervertebral disc (IVD) degeneration is thought to play a major role in chronic back and neck pain. Decades of bench-top research in tissue mechanics have shown clear relationships between changes in mechanical properties and abnormal changes IVD structure and composition. Our overall hypothesis is that measurements of IVD mechanical properties can provide valuable information about its structure and composition for early diagnosis of degeneration, quantification of degeneration progress, and evaluation of treatment strategies. Magnetic Resonance Elastography (MRE) is an imaging method to quantify mechanical properties from soft tissues. The objectives of this study are to evaluating repeatability and collecting base line data from healthy individuals; and to apply MRE to patients with disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy controls must be generally healthy individuals in the age range of 18-65.
* Patients, 18 to 65 years old, who have undergone or will undergo MRI as part of the diagnosis of back pain and are diagnosed with one or more herniated discs in the lumbar spine (aka, disc rupture).

Exclusion Criteria:

* Participants with a history of neurological injury or disease will be excluded.
* Participants with contraindications to MRI scanning will be excluded (e.g., electric/mechanical implant, device such as a pacemaker).
* Participants who are claustrophobic will be excluded.
* Participants who are >250 lbs will be excluded (due to weight and physical constraints of - the scanner, i.e., 55 cm bore).
* Those unable to consent, pregnant women, children, and prisoners will be excluded.
* People under the age of 18 will be excluded as well.
* Individuals who do not understand English (written or spoken) will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in mechanical properties of the herniated intervertebral disc | 1 week
  It is expected that MR Elastography can measure changes in mechanical properties of the herniated intervertebral disc.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Cortes, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No